CLINICAL TRIAL: NCT05846646
Title: Phase 2 Randomized Clinical Trial Comparing the Safety and Efficacy of PULSAR-Integrated Radiotherapy + Pembrolizumab or Nivolumab Administered With or Without STING-Agonist IMSA101 in Patients With Oligometastatic NSCLC and RCC
Brief Title: Study of PULSAR-ICI +/- IMSA101 in Patients With Oligometastatic NSCLC and RCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in ImmuneSensor corporate strategy.
Sponsor: ImmuneSensor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMSA101-102
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Oligometastatic Disease
Keywords: Non-small cell lung cancer (NSCLC); Renal cell carcinoma (RCC); Adult
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — Immune Checkpoint Inhibitors; pembrolizumab; Nivolumab; DEAE-Dextran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): PULSAR-ICI + IMSA101
  Interventions: Drug: IMSA101; Drug: Immune checkpoint inhibitor; Radiation: PULSAR
- Control Arm (Active Comparator): PULSAR-ICI
  Interventions: Drug: Immune checkpoint inhibitor; Radiation: PULSAR

INTERVENTIONS:
Drug: IMSA101 — Intra-tumoral administration once weekly for the first three weeks of Cycle 1 (Days 1, 8 and 15) and then on Day 1 of Cycles 2 and 3.
  Arms: Experimental Arm
Drug: Immune checkpoint inhibitor — 1st infusion on Cycle 1 Day 2, and then thereafter as per product label
  Other Names: pembrolizumab; nivolumab
Radiation: PULSAR — 1st day of Cycles 1, 2 and 3.

SUMMARY:
Phase 2, open-label, multicenter, randomized study comparing the safety and efficacy of personalized ultra-fractionated stereotactic adaptive radiotherapy (PULSAR) combined with immune checkpoint inhibitor (ICI) immunotherapy (PULSAR-ICI) + IMSA101 and PULSAR-ICI alone in patients with NSCLC or RCC

DETAILED DESCRIPTION:
Patients shall be enrolled in 2 treatment arms as follows:

1. 20 patients in the control arm (PULSAR-ICI alone)
2. 20 patients in the experimental arm (PULSAR-ICI + IMSA101)

Patients will be stratified by histology (NSCLC and RCC) in the randomized portion.

PULSAR-ICI with or without IMSA101 treatment will be administered to the patients in Cycles 1, 2, and 3, and thereafter only standard of care ICI monotherapy will be administered to all patients. Each treatment cycle will be 28 days in duration for Cycles 1, 2 and 3, then per standard of care monotherapy thereafter based on the product labels of the prescribed ICI.

The study will start with a safety run-in portion at 2 dose levels for the experimental arm, followed by a randomized portion for both treatment arms. The safety run-in shall employ a 3+3 safety run-in component.

All patients will be followed throughout the study for drug tolerability and safety by collecting clinical and laboratory data, including adverse events (AEs) using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 criteria, SAEs, concomitant medications, and vital signs.

All patients will be assessed for anti-tumor efficacy at screening, prior to the end of Cycle 3, and at 8-week intervals thereafter based on radiographic assessments (all outcome measures per RECIST Version 1.1 and iRECIST).

All patients will continue to receive their assigned treatment throughout the study until the occurrence of disease progression (based on iRECIST), death, or other unacceptable treatment-related toxicity, or until the study is closed by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Signed informed consent and mental capability to understand the informed consent
3. Histologically or cytologically documented NSCLC or RCC with radiographically documented presence of ≤ 6 metastatic lesions consistent with the diagnosis of "oligometastatic" disease
4. Patient's disease must be evaluable per RECIST Version 1.1
5. All metastatic lesions amenable to administration of radiotherapy, at the discretion of the investigator
6. Must have at least one single pre-defined lesion/lesion site (longest diameter ≥ 10 mm and ≤ 50 mm) suitable for intra-tumoral injection
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
8. Electrocardiogram (ECG) without evidence of clinically significant conduction abnormalities or active ischemia as determined by the investigator
9. Acceptable organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) > 1,500 cells/μL
   * Platelets > 50,000 cells/μL
   * Total bilirubin ≤ 1.5 times (×) the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN. If liver metastases are present, AST/ALT < 5 × ULN
   * Serum creatinine < 1.5 mg/dL and a measured creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault formula
   * Prothrombin time (PT)/partial thromboplastin time (PTT) ≤ 1.5 × ULN
10. Women of child-bearing potential (defined as a female who has experienced menarche and who has not undergone successful surgical sterilization [hysterectomy, bilateral salpingectomy, or bilateral oophorectomy]) or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months with an appropriate clinical profile at the appropriate age, eg, greater than 45 years) must have a negative serum pregnancy test prior to first dose of study treatment
11. Male and female patients with reproductive potential must agree to use two forms of highly effective contraception throughout the study

Exclusion Criteria:

1. Prior disease progression through programmed cell death ligand 1 (PD-L1 or PD-1)-targeted immunotherapy
2. Prior receipt of stimulator of interferon genes (STING) agonist
3. Prior receipt of therapeutic radiotherapy to the lesions intended for PULSAR treatment
4. Anti-cancer therapy, except pembrolizumab and nivolumab, within 4 weeks or < 5 half-lives of the first dose of study treatment
5. Existence of primary tumor that requires therapeutic treatment beyond the provided immune checkpoint inhibitor drug
6. Failure to recover, to Grade 1 or less, from clinically significant AEs due to prior anti-cancer therapy, as judged by the investigator
7. Previous life-threatening (Grade 4) immune-related adverse event (irAE)
8. Existence of actionable mutations that may be eligible for mutation-targeted drug that represents standard-of-care therapy
9. Presence of brain metastases
10. Baseline prolongation of QT/corrected QT (QTc) interval (QTc interval > 470)
11. Uncontrolled intercurrent illness (including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations) that in the opinion of the investigator would limit compliance with study requirements
12. Women who are pregnant or breastfeeding
13. Sponsor reserves the right to exclude any patient from the study on the basis of pre-study medical histories, physical examination findings, clinical laboratory results, prior medications, or other entrance criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Widhelm, Study Director — ImmuneSensor Therapeutics
Locations (9):
- United States (9):
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated early by sponsor due to change in corporate strategy.
Groups:
- Experimental Arm (800 mcg): PULSAR-ICI + IMSA101 (800 mcg)
- Experimental Arm (1200 mcg): PULSAR-ICI + IMSA101 (1200 mcg)
- Control Arm: PULSAR - ICI
Period: Overall Study
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Started | 3 | 3 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Early Study Termination | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled to Safety Run In portion of trial where all everyone assigned to Experimental Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm | Total
Number analyzed (Participants) | 3 | 3 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 1
  >=65 years | 3 | 2 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 0 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Effects
Description: Progression-free rate at 18 months
Time Frame: 18 months
Population: Data were not collected due to study termination prior to participants' assessment at the 18-month time point
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Occurrence of treatment-related adverse events
Time Frame: Enrolment through end of study period (1 year, 3 months). AE data captured continually.
Population: Zero patients enrolled to Control Arm during Safety Run In period.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Arm (1200 mcg): PULSAR-ICI + IMSA101 (1200 mcg
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Number analyzed (Participants) | 3 | 3 | 0
Participants | 3 | 3 | 0

3. Secondary Outcome: Anti-tumor Effects
Description: Progression-free at 8-week intervals from 6 months to 22 months
Time Frame: 6 to 22 months
Population: Data were not collected due to study termination prior to participants' assessment at the 18-month time point
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Anti-tumor Effects
Description: Time to progression
Time Frame: upon enrolment through end of study period (2 years)
Population: Data were not collected due to study termination prior to participants' assessment at the 18-month time point
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Anti-tumor Effects
Description: Overall response rate, duration of response, progression-free survival
Time Frame: upon enrolment through end of study period (2 years)
Population: Data were not collected due to study termination prior to participants' assessment at the 18-month time point
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Quality of Life (QoL)
Description: Patient reported outcome on FACT-G questionnaire
Time Frame: upon enrolment through end of study period (2 years)
Population: Data were not collected due to study termination prior to participants' assessment at the 18-month time point
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrolment through end of study period (1 year, 3 months). AE data captured continually.
Description: Analysis population is the six patients enrolled to the Experimental Arm.
Arm/Group | Experimental Arm (800 mcg) | Experimental Arm (1200 mcg) | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (800 mcg) (N=3) | Experimental Arm (1200 mcg) (N=3) | Control Arm (N=0)
Possible Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (800 mcg) (N=3) | Experimental Arm (1200 mcg) (N=3) | Control Arm (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 3 | 2 | 0
Fatigue (General disorders) | 2 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Pain (General disorders) | 0 | 2 | NA
Pyrexia (General disorders) | 1 | 1 | 0
Weight decreased (Investigations) | 2 | 1 | 0
Decreased Appetite (Investigations) | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Study terminated early due to change in ImmuneSensor strategic direction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT05846646/Prot_SAP_000.pdf